CLINICAL TRIAL: NCT00240188
Title: Ventral Incisional Hernia Repair: Comparison Of Laparoscopic and Open Repair With Mesh
Brief Title: A Study to Compare Ventral Incisional Hernia by Laparoscopic vs Open Repair With Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Itani, Kamal - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-011-03S
Record Dates: First submitted 2005-08-30; First posted 2005-10-17 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Hernia, Ventral
Keywords: Hernia; Incisional; Laparoscopic; Mesh; Repair; Ventral
MeSH Terms: conditions — Hernia, Ventral; Hernia; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Open mesh repair of ventral incisional hernia; Procedure: Laparoscopic mesh repair of ventral incisional hernia

INTERVENTIONS:
Procedure: Open mesh repair of ventral incisional hernia — For the open procedure, the technique, as described by Chevrel and others was adopted.
Procedure: Laparoscopic mesh repair of ventral incisional hernia — For the laparoscopic repair, the method of Gagner was adopted

SUMMARY:
The purpose of this research is to compare open ventral incisional hernia repair to the laparoscopic repair with respect to complications, recurrence, pain, return to normal activities of daily living, and return to work.

DETAILED DESCRIPTION:
The appearance of ventral incisional hernia (VIH) following an open abdominal operation is an important postoperative problem. While advances in anesthesia techniques, better methods to prevent surgical infections, and improved treatment of infection, and the use of new suture materials have reduced the incidence of incisional hernias, incisional hernias still occurs in 0.5-11% of all open abdominal surgical procedures performed.

Overview of study design: We are conducting a 4 center randomized clinical trial to compare the outcomes of two methods of surgical management of ventral incisional hernia. Patients presenting to a physician with a ventral incisional hernia will be considered for the trial. The study is designed to compare the rate of complications, pain, time to return to normal activities, Health related quality of life (HRQoL) and patient satisfaction between laparoscopic and open mesh repair for ventral incisional hernia. The rate of recurrence of the hernia at 1-2 years will be evaluated as a secondary outcome. Four VA medical centers with the capability of enrolling 40-50 patients a year have been selected based on volume, experience with open and laparoscopic ventral herniorrhaphy and experience in the conduct of clinical trials. Patients are recruited by physicians at each site and referred to the site coordinator who screens them for eligibility. The trial is randomized but not blinded. The randomization scheme takes into consideration that random allocation of patients to each study group is made within each center. In addition to the participating center, the other baseline variables that serve as stratification factors are first time or recurrent ventral incisional hernia and patient with a body mass index greater or less than 35arm.

Timeline: The trial consists of 3 phases: Implementation, Patient intake and follow-up, closeout and final analysis. 1-Implementation (2 months): The implementation which will include funding, recruitment of the nurse coordinators and review of the study protocol and techniques of operation was 2 months in duration. 2-Patient intake and follow up (32 months): All study patients are recruited during that period of time. Follow-up will occur simultaneously and will end at close out. The range of follow-up is expected to range from 8 weeks to 34 months. 4-Final analysis and closeout: The participating centers will be given 2 months of funding to close out the data collection. During this period, all final follow-up visits and data collection will be completed. Final analysis will run concurrently with closeout.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for enrollment into the study if they meet the following criteria: -Are 18 years of age or older -Have a diagnosis of ventral primary incisional hernia 9-225 cm2 in size. -Give informed consent for randomization - Have a negative pregnancy test. (Women)

Exclusion Criteria:

Patients will be excluded for the following reasons: -Hernia cannot be detected on physical examination - Primary ventral or umbilical hernia - Small hernia defined as less than 9 cm2 - Giant hernia defined as greater than 225 cm2 in size - ASA class 4 or 5, or contraindications to general anesthesia - Severe co morbid conditions likely to limit survival to less than 3 years - History of malignancy within the past 5 years except for non-melanoma skin cancer - Cirrhosis with or without ascites - Presence of bowel obstruction( partial or intermittent), strangulation, peritonitis, or perforation. - Presence of local or systemic infection - Participation in another clinical trial - Emergency operation - Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Overall complication rates at eight weeks and the odds of complications, adjusted for study site, body mass index, and hernia type | Eight (8) weeks post-operatively

SECONDARY OUTCOMES:
Compare pain, return to normal activities of daily living, and return to work. Health related quality of life, and recurrence. | One (1) and two (2) years post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Itani, MD, Principal Investigator — VA Boston Healthcare System, Boston
Locations (1):
- VA Boston Healthcare System, Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Kaafarani HM, Hur K, Campasano M, Reda DJ, Itani KM. Classification and valuation of postoperative complications in a randomized trial of open versus laparoscopic ventral herniorrhaphy. Hernia. 2010 Jun;14(3):231-5. doi: 10.1007/s10029-009-0593-z. Epub 2010 Mar 6. PMID 20213456
- [Result] Kaafarani HM, Kaufman D, Reda D, Itani KM. Predictors of surgical site infection in laparoscopic and open ventral incisional herniorrhaphy. J Surg Res. 2010 Oct;163(2):229-34. doi: 10.1016/j.jss.2010.03.019. Epub 2010 Apr 1. PMID 20605590
- [Result] Itani KM, Neumayer L, Reda D, Kim L, Anthony T. Repair of ventral incisional hernia: the design of a randomized trial to compare open and laparoscopic surgical techniques. Am J Surg. 2004 Dec;188(6A Suppl):22S-29S. doi: 10.1016/j.amjsurg.2004.09.006. PMID 15610889
- [Result] Kaafarani HM, Hur K, Hirter A, Kim LT, Thomas A, Berger DH, Reda D, Itani KM. Seroma in ventral incisional herniorrhaphy: incidence, predictors and outcome. Am J Surg. 2009 Nov;198(5):639-44. doi: 10.1016/j.amjsurg.2009.07.019. PMID 19887192
- [Result] Itani KM, Hur K, Kim LT, Anthony T, Berger DH, Reda D, Neumayer L; Veterans Affairs Ventral Incisional Hernia Investigators. Comparison of laparoscopic and open repair with mesh for the treatment of ventral incisional hernia: a randomized trial. Arch Surg. 2010 Apr;145(4):322-8; discussion 328. doi: 10.1001/archsurg.2010.18. PMID 20404280